CLINICAL TRIAL: NCT00599768
Title: Development and Validation for Taiwan Version ID Pain Questionnaire (ID Pain-T) and DN4 Questionnaire.
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A0081175; TWN-2006-CNS-001
Record Dates: First submitted 2008-01-11; First posted 2008-01-24 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2009-11

CONDITIONS: Neuralgia; Nerve Pain; Neuropathic Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: ID-Pain DN4 Questionnaire — This is a non-interventional questionnaire validation study

SUMMARY:
This prospective cohort and multi-site study aims to develop Taiwan version (ID Pain-T) based on the original versions of ID Pain and also DN4, and validate both ID Pain-T and DN4 applied in Taiwanese subjects at the clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Subjects without headache pain over 30 days and at least 18 years old who will visit the clinic, inclusive of male and female.
* Subjects who are able to complete the ID Pain-T Questionnaire.

Exclusion Criteria:

* Subjects who are illiterate or unable to complete questionnaire.
* Subjects who are currently participating in another study or have participated in another pain study within one month of study entry.
* Subjects with low back pain are unable to participate in this study; as the sciatica caused by the piriformis (exclusive of the other types of sciatic pain), lumbago, unclear identification in nerve injury (e.g. complex regional pain syndrome type I) or mixed origin (e.g. cancer pain).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients of non-headache pain for more than 30 days and those whose age is more than 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 325 (Actual)
Dates: Start 2008-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Determine the optimal cut-off score of ID Pain-T Questionnaire for screening of neuropathic pain | end of study

SECONDARY OUTCOMES:
Evaluate the predictive power of ID Pain-T Questionnaire for diagnosis of neuropathic pain | end of study
Develop and evaluate validity of a short form diagnostic tool based on DN4 structure | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081175&StudyName=Development%20and%20Validation%20for%20Taiwan%20Version%20ID%20Pain%20Questionnaire%20%28ID%20Pain-T%29%20and%20DN4%20Questionnaire.